CLINICAL TRIAL: NCT02393209
Title: A Phase 1b/Adaptive Phase 2 Study of Docetaxel With or Without MLN1117 in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Docetaxel With or Without TAK-117 (MLN1117) in Participants With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy in combination.
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLN1117-1501; 2014-004281-25 (EudraCT Number); U1111-1160-1736 (Registry Identifier: UTN (WHO))
Record Dates: First submitted 2015-03-15; First posted 2015-03-19 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Drug therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; serabelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TAK-117 200 mg + Docetaxel (36 mg/m^2) (Experimental): TAK-117 200 mg, tablets, orally on Days 2, 3, 4, 9, 10, 11, 16, 17, and 18 of the 21-day cycle and docetaxel 36 mg/m^2, intravenous (IV) infusion, on Days 1 and 8 of the 21-day cycle up ro Cycle 9 (approximately 189 days).
  Interventions: Drug: Docetaxel; Drug: TAK-117
- TAK-117 300 mg + Docetaxel 36 mg/m^2 (Experimental): TAK-117 200 mg, tablets, orally on Days 2, 3, 4, 9, 10, 11, 16, 17, and 18 of the 21-day cycle and docetaxel 36 mg/m^2, IV infusion, on Days 1 and 8 of the 21-day cycle up to 6 cycles (approximately 126 days).
  Interventions: Drug: Docetaxel; Drug: TAK-117
- Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 (Experimental): TAK-117 tablets, at the dose determined in the dose escalation phase, on Days 2, 3, 4, 9, 10, 11, 16, 17, and 18 of a 21-day cycle plus Docetaxel 36 mg/m^2 IV infusion on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Docetaxel; Drug: TAK-117
- Phase 2 - Docetaxel 75 mg/m^2 (Experimental): Docetaxel 75 mg/m^2, IV infusion once every 3 weeks (per approved prescribing information) with dosing on Day 1 of each 21-day cycle.
  Interventions: Drug: Docetaxel; Drug: TAK-117

INTERVENTIONS:
Drug: Docetaxel — Docetaxel intravenous infusion
Drug: TAK-117 — TAK-117 Tablets
  Other Names: MLN1117

SUMMARY:
The purpose of this study is to determine the recommended phase 2 dose (RP2D) of TAK-117 when administered in combination with docetaxel in participants with non-small cell lung cancer (NSCLC) and to evaluate efficacy, safety, and tolerability of TAK-117 administered alone and in combination with docetaxel at the RP2D in participants with locally advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
The drug being evaluated in this study is called TAK-117. TAK-117 is tested in combination with docetaxel versus docetaxel alone for the treatment of non-small cell lung cancer (NSCLC).

This study consisted of 2 phases:

* Phase 1b - dose escalation phase
* Phase 2 - expansion phase.

The study enrolled 14 patients with NSCLC who have been treated with multiple prior lines of therapies will be enrolled for Phase 1b. The participants will receive docetaxel (36 mg/m^2) intravenous (IV) and TAK-117 tablets, orally administered, once daily in 21-day dosing cycles. The TAK-117 dose will be escalated until recommended Phase 2 dose (RP2D) is determined.

Each part of the adaptive Phase 2 portion of the study is designed as a stand-alone, randomized study evaluating PFS as the primary efficacy measure in a total of 60 participants between the 2 treatment arms: TAK-117 plus docetaxel versus docetaxel alone. An event-driven analysis of PFS will be performed after each part of Phase 2. On the basis of the PFS analysis of the preceding part of the study, the study may be stopped for efficacy or futility, or proceed to the next part. However, Phase 2 of the study was cancelled.

Study drug will be administered in 21-day dosing cycles. During each phase of the study, participants will be treated with a maximum of 9 cycles of either docetaxel alone or docetaxel plus TAK-117. Subsequently, participants treated with docetaxel plus TAK-117 may continue to receive TAK-117 monotherapy until progression of disease, occurrence of unacceptable toxicities or death.

The maximum duration of treatment for participants will be 12 months unless it is determined that a participant would derive benefit from continued treatment beyond 12 months. Participants will continue to be followed after discontinuation of study drug to collect PFS and OS data. Participants may withdraw from therapy at any time.

This multicenter trial will be conducted in North America. The overall time to participate in this study is up to 24 months.

ELIGIBILITY:
Inclusion Criteria

* Has a histologically and/or cytologically confirmed diagnosis of NSCLC (squamous or nonsquamous).

  - For Phase 2 of the study, has a diagnosis of mixed squamous and nonsquamous (or adenosquamous) NSLC.
* Has locally advanced or metastatic disease (Stage IIIb or Stage IV) with radiographically or clinically evaluable lesions.
* Has experienced failure of at least 1 prior chemotherapy regimen:

  * For Phase 2 of the study:
  * Participants must have received 1 prior platinum-based chemotherapy regimen (excluding a docetaxel-containing regimen) for advanced or metastatic (Stage IIIb or Stage IV) disease followed by documented progressive disease (PD).
  * A drug provided as maintenance therapy following cytotoxic chemotherapy will be considered to be part of that regimen.
  * Participants who received prior therapy with paclitaxel as a part of the platinum-based doublet front-line regimen without PD on therapy.
  * Participants who, after the front-line, platinum-based, non-docetaxel containing chemotherapy, have been treated with 1 line of nivolumab or other immune-checkpoint inhibitors but progressed on or after the therapy.
  * For Phase 1b of the study: Participants who have experienced failure of multiple lines of prior chemotherapy are eligible.
  * For Phase 2, has archived or fresh tumor biopsy samples (obtained during screening) sufficient for genotyping.
* Has adequate organ function, before the first dose of study drug.
* Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Female participants who are postmenopausal for at least 1 year before the screening visit or are surgically sterile, or are of childbearing potential, agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 30 days (or longer, as mandated by local labeling) after the last dose of study drug, or agree to practice true abstinence.
* Female participants must agree to not donate eggs (ova) during the course of this study and for 30 days after receiving their last dose of TAK-117 and, for docetaxel, for as long as is mandated by local labeling.
* Male participants agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of TAK-117 and, for docetaxel, for as long as is mandated by local labeling, or agree to practice true abstinence.
* Male participants must agree to not donate sperm during the course of the study and for 120 days after receiving their last dose of TAK-117 and, for docetaxel, for as long as is mandated by local labeling.
* Has suitable venous access for the study-required blood sampling.
* Has recovered (ie, <= Grade 1 toxicity or eligibility per this protocol is met) from the reversible effects of prior anticancer therapy.
* In the opinion of the investigator, the participant or legal guardian is capable of understanding and complying with protocol requirements for the duration of the study.

Exclusion Criteria:

* Previous treatment with a PI3K or AKT inhibitor.
* Prior cancer therapy or other investigational therapy within 2 weeks before the first administration of study drug or failed to recover from the reversible effects of prior anticancer therapies. For prior therapies with a half-life longer than 3 days, the interval must be at least 28 days before the first administration of study drug, and the participant must have documented progressive disease.
* Has poorly controlled diabetes mellitus defined as HbA1c > 6.5%.
* Has taken strong inhibitors or strong inducers of CYP3A4 within 14 days before the first dose of study drug.
* Has taken histamine-H2 receptor antagonists and/or neutralizing antacids within 24 hours before the first administration of study drug.
* Has taken proton pump inhibitors within 7 days before the first administration of study drug.
* Has a condition that requires the concomitant use of any of the protocol-excluded medications, supplements, or food products during the course of the study .
* Has any clinically significant co-morbidities.
* Has acute myocardial infarction within 6 months before starting study drug, current or history of New York Heart Association Class III or IV heart failure; evidence of current uncontrolled cardiovascular conditions including cardiac arrhythmias, angina, pulmonary hypertension, or electrocardiogram (ECG) evidence of acute ischemia or active conduction system abnormalities; Fridericia's corrected QT interval > 475 milliseconds (msec) (males) or > 450 msec (females) on a 12-lead ECG during the Screening period; or abnormalities on 12-lead ECG including, but not limited to, changes in rhythm and intervals that in the opinion of the investigator are considered to be clinically significant.
* Has known, previously diagnosed human immunodeficiency virus infection or active chronic hepatitis B or C.
* Has brain metastasis, unless has completed definitive therapy, is not on steroids, has a stable neurologic status for at least 2 weeks after completion of the definitive therapy and steroids, and does not have neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Has active secondary malignancy that requires treatment.
* Has any serious medical or psychiatric illness, including drug or alcohol abuse.
* Male participants who intend to donate sperm during the course of this study or 120 days after receiving their last dose of TAK-117 and, for docetaxel, for as long as is mandated by local labeling.
* Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 before administration of the first dose of study drug.
* Is unwilling or unable to abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (11):
- United States (6):
  - San Diego, California
  - Atlanta, Georgia
  - Farmington Hills, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Chattanooga, Tennessee
- Canada (2):
  - Edmonton, Alberta
  - Toronto, Ontario
- Netherlands (3):
  - Amsterdam
  - Hoofddorp
  - Maastricht

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in United States and 1 in Canada from 03 June 2015 to 20 January 2017. The Phase 2 portion of the study was cancelled by the sponsor.
Pre-assignment Details: Participants with a diagnosis of metastatic non-small lung cancer were enrolled in a dose escalation study and received one of 2 doses: TAK-117 (200 mg) plus docetaxel or TAK-117 (300 mg) plus docetaxel.
Groups:
- Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2: TAK-117 200 mg, tablets, orally on Days 2, 3, 4, 9, 10, 11, 16, 17, and 18 of the 21-day cycle and docetaxel 36 mg/m^2, intravenous (IV) infusion, on Days 1 and 8 of the 21-day cycle up to 9 cycles (approximately 189 days).
- Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2: TAK-117 300 mg, tablets, orally on Days 2, 3, 4, 9, 10, 11, 16, 17, and 18 of the 21-day cycle and docetaxel 36 mg/m^2, IV infusion, on Days 1 and 8 of the 21-day cycle up to 6 cycles (approximately 126 days).
Period: Overall Study
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2 | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Started | 6 | 8 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 8 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 1 | 0 | 0
Not completed — Withdrawal by Patient | 1 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 0 | 0
Not completed — Death due to Disease Progression | 2 | 2 | 0 | 0
Not completed — Death from Legionella Infection | 0 | 1 | 0 | 0
Not completed — Patient Seen by Another Oncologist | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed for enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2 | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.10) | 62.1 (11.32) | 62.9 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 7 | 12
  Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 9
  Black or African American | 1 | 2 | 3
  Asian | 1 | 0 | 1
  Not reported | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 171.53 (5.854) | 172.95 (6.102) | 172.34 (5.810)
Weight [Mean (Standard Deviation); unit: kg] | 69.48 (21.630) | 72.69 (9.157) | 71.31 (15.093)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body Surface Area (m^2) = Square root [height (cm) * weight (kg) / 3600].
  m^2 | 1.805 (0.2987) | 1.865 (0.1231) | 1.839 (0.2084)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT) in Phase 1b
Description: DLT was evaluated according to National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 and was defined as any of the following events: 1. Grade 4 neutropenia or thrombocytopenia lasting ≥7 consecutive days; 2. Grade 4 neutropenia with fever and/or infection; 3. Platelet count <10,000/mm^3; 4. ≥Grade 3 thrombocytopenia with bleeding; 5. Any other ≥Grade 4 hematologic toxicity; 6. Any other ≥Grade 3 nonhematologic toxicity, with following exceptions: ≥Grade 3 arthralgia/myalgia, ≥Grade 3 nausea/emesis, ≥Grade 3 diarrhoea, Grade 3 fatigue, Grade 3 Rash, Grade 3 nonhematological toxicity that could be controlled to ≤Grade 1 with appropriate treatment; 7. Inability to administer at least 75% of planned doses; 8. Clinically significant occurrence per investigator that is a safety risk.
Time Frame: Cycle 1 (Up to Day 21)
Population: The DLT-evaluable population was defined as all participants who either experienced DLT during Cycle 1 or complete treatment with at least 75% of the planned doses of TAK-117 plus docetaxel and have sufficient follow-up data to allow investigators and sponsor to determine whether DLT occurred.
Measure: Number; unit: participants
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 6 | 8
participants | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD) of TAK-117 in Combination With Docetaxel 36 mg/m^2 in Phase 1b
Description: The MTD is defined as the dose of TAK-117 in combination with docetaxel 36 mg/m^2 at which 1 of 6 evaluable participants experience DLT. DLT was evaluated according to NCI CTCAE version 4.03 and was defined as any of the following events: 1. Grade 4 neutropenia or thrombocytopenia lasting ≥7 consecutive days; 2. Grade 4 neutropenia with fever and/or infection; 3. Platelet count <10,000/mm^3; 4. ≥Grade 3 thrombocytopenia with bleeding; 5. Any other ≥Grade 4 hematologic toxicity; 6. Any other ≥Grade 3 nonhematologic toxicity, with following exceptions: ≥Grade 3 arthralgia/myalgia, ≥Grade 3 nausea/emesis, ≥Grade 3 diarrhoea, Grade 3 fatigue, Grade 3 Rash, Grade 3 nonhematological toxicity that could be controlled to ≤Grade 1 with appropriate treatment; 7. Inability to administer at least 75% of planned doses; 8. Clinically significant occurrence per investigator that is a safety risk.
Time Frame: Cycle 1 (Up to Day 21)
Population: as for outcome 1
Measure: Number; unit: mg
Groups:
- TAK-117 + Docetaxel: TAK-117 200 mg or 300 mg, tablets, orally on Days 2, 3, 4, 9, 10, 11, 16, 17, and 18 of the 21-day cycle and docetaxel 36 mg/m^2, IV infusion, on Days 1 and 8 of the 21-day cycle up to 9 cycles (approximately 189 days).
Arm/Group | TAK-117 + Docetaxel
Number analyzed (Participants) | 14
mg | 300

3. Primary Outcome: Recommended Phase 2 Dose of TAK-117 in Phase 1b
Description: The recommended phase 2 dose was determined in Phase 1b based on participant dose-limiting toxicities and the maximum tolerated dose.
Time Frame: Cycle 1 (Up to Day 21)
Population: as for outcome 1
Measure: Number; unit: mg
Arm/Group | TAK-117 + Docetaxel
Number analyzed (Participants) | 14
mg | 200

4. Primary Outcome: Progression-Free Survival (PFS) in Phase 2
Description: PFS is defined as the time from the date randomization to the date of first documented progressive disease (PD) or death as assessed by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. PD is defined as 20% increase in the sum of the longest diameter of target lesions for measurable neoplastic disease.
Time Frame: Approximately 12 months in Phase 2
Population: Data was not analyzed as Phase 2 of the study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Significant Change in Vital Signs Reported as Adverse Events in Phase 1b
Description: Clinically significant change from baseline in vital sign measures will be assessed. Vital sign measurements included measurements of diastolic and systolic blood pressure, heart rate, and temperature.
Time Frame: First dose of study drug through 30 days after the last dose of study drug (Up to Day 223)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 6 | 8
participants
  Bradycardia | 1 | 0
  Sinus tachycardia | 0 | 1

6. Secondary Outcome: Number of Participants With Significant Change in Physical Examination Reported as Adverse Events in Phase 1b
Description: Physical examination consists of examinations of the following body systems: (1) eyes; (2) ears, nose, throat; (3) cardiovascular system; (4) respiratory system; (5) gastrointestinal system; (6) dermatologic system; (7) extremities; (8) musculoskeletal system; (9) nervous system; (10) lymph nodes; and (11) physical examinations other than body systems described in (1) to (10).
Time Frame: First dose of study drug through 30 days after the last dose of study drug (Up to Day 223)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 6 | 8
participants | 0 | 1

7. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings Reported as Adverse Events in Phase 1b
Description: A standard 12-lead ECG was performed.
Time Frame: First dose of study drug through 30 days after the last dose of study drug (Up to Day 223)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 6 | 8
participants
  Bradycardia | 1 | 0
  Tachycardia | 0 | 1

8. Secondary Outcome: Number of Participants With Clinically Significant Change in Clinical Laboratory Tests Reported as Adverse Events in Phase 1b
Description: The number of participants with any markedly abnormal standard safety laboratory values (Chemistry, Hematology and Urinalysis) collected throughout study.
Time Frame: First dose of study drug through 30 days after the last dose of study drug (Up to Day 223)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 6 | 8
participants
  Anemia | 2 | 2
  Hypokalemia | 1 | 3
  Hypomagnesemia | 0 | 3
  Hypophosphatemia | 0 | 3
  Aspartate aminotransferase increased | 1 | 2
  Febrile neutropenia | 1 | 2
  Hyponatremia | 1 | 2
  Hyperglycemia | 0 | 2
  Leukopenia | 0 | 1
  Pancytopenia | 0 | 1
  Thrombocytopenia | 1 | 0
  Blood creatinine increased | 1 | 1
  Alanine aminotransferase increased | 0 | 1
  Blood cholesterol increased | 0 | 1
  Neutrophil count decreased | 1 | 0
  White blood cell count decreased | 0 | 1
  Hyperkalaemia | 1 | 0
  Hypernatraemia | 0 | 1
  Hypoalbuminaemia | 1 | 0
  Hypocalcaemia | 0 | 1

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) in Phase 1b
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug to 30 days after last dose of study drug (Up to Day 223)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 6 | 8
participants
  TEAEs | 6 | 8
  SAEs | 5 | 6

10. Secondary Outcome: Number of Participants With Significant Change in Vital Signs Reported as Adverse Events in Phase 2
Description: Vital signs (blood pressure, pulse rate, and oral temperature) measurements were collected throughout the study.
Time Frame: Approximately 12 months in Phase 2
Population: Data was not analyzed as Phase 2 of study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With Significant Change in Physical Examination Reported as Adverse Events in Phase 2
Description: as for outcome 6
Time Frame: Approximately 12 months in Phase 2
Population: Data was not analyzed as Phase 2 of study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Findings Reported as Adverse Events in Phase 2
Description: Clinically significant changes from baseline in ECGs will be tabulated by time point including any unscheduled measurements.
Time Frame: Approximately 12 months in Phase 2
Population: Data was not analyzed as Phase 2 of study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Change in Clinical Laboratory Tests Reported as Adverse Events in Phase 2
Description: as for outcome 8
Time Frame: Approximately 12 months in Phase 2
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) in Phase 2
Description: as for outcome 9
Time Frame: Approximately 12 months in Phase 2
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Response Rate in Phase 2
Description: Response rate is defined as the percentage of participants with Complete Response (CR) + Partial Response (PR) as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1. According to RECIST: CR is defined as disappearance of all target lesions and PR is defined as 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Approximately 12 months in Phase 2
Population: Data was not analyzed as Phase 2 of the study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Disease Control Rate in Phase 2
Description: Disease control rate is defined as percentage of participants with CR + PR + stable disease (SD). According to RECIST: CR is defined as disappearance of all target lesions, PR is defined as 30% decrease in the sum of the longest diameter of target lesions and SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter (LD) since the treatment started.
Time Frame: Approximately 12 months in Phase 2
Population: Data was not analyzed as Phase 2 of the study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Duration of Response in Phase 2
Description: The duration of response is defined as the time from the date of first documentation of a response to the date of first documentation of progression of disease. As per RECIST 1.1, PD is defined as 20% increase in the sum of the longest diameter of target lesions for measurable neoplastic disease.
Time Frame: Approximately 12 months in Phase 2
Population: Data was not analyzed as Phase 2 of the study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Time to Progression in Phase 2
Description: Time to progression is defined as the time from the date of randomization to the date of first documentation of progression of disease. As per RECIST 1.1, PD is defined as 20% increase in the sum of the longest diameter of target lesions for measurable neoplastic disease.
Time Frame: Approximately 12 months in Phase 2
Population: Data was not analyzed as Phase 2 of the study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Overall Survival (OS) in Phase 2
Description: Overall survival is defined as the time from the date of randomization to the date of death.
Time Frame: Approximately 12 months in Phase 2
Population: Data was not analyzed as Phase 2 of the study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: TAK-117 Plasma Concentration in Phase 1b
Time Frame: Cycle 1 Day 1 pre-dose and 0.5, 1, 2, 4, 6, 8 and 24 hours post-dose
Population: The PK-evaluable population was defined as all participants for whom there are sufficient dosing and TAK-117 concentration-time data to permit non-compartmental PK analysis. Here 'Number Analyzed' are participants analyzed at the specific timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 6 | 7
ng/mL
  Predose: number analyzed (Participants) | 5 | 7
  Predose | 114.00 (254.912) | 0.00 (0.000)
  0.5 Hour Postdose: number analyzed (Participants) | 5 | 7
  0.5 Hour Postdose | 1208.60 (1080.782) | 847.39 (966.346)
  1 Hour Postdose | 1907.00 (1307.124) | 1973.29 (1688.210)
  2 Hours Postdose | 2597.83 (1612.233) | 3021.43 (2162.417)
  4 Hours Postdose | 2477.50 (1407.465) | 4185.71 (2156.439)
  6 Hours Postdose: number analyzed (Participants) | 5 | 7
  6 Hours Postdose | 2143.00 (1290.395) | 3648.57 (1636.892)
  8 Hours Postdose | 1902.50 (1210.553) | 3677.14 (1941.020)
  24 Hours Postdose | 652.17 (472.315) | 1771.57 (1347.864)

21. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-117
Time Frame: Cycle 1 Day 1 pre-dose and 0.5, 1, 2, 4, 6, 8 and 24 hours post-dose
Population: This analysis was not performed due to lack of data.
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-117
Time Frame: Cycle 1 Day 1 pre-dose and up to 24 hours post-dose
Population: This analysis was not performed due to lack of data.
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: AUCtau: Area Under the Concentration Time Curve From Time 0 to the Next Dose in Phase 1b for TAK-117
Time Frame: Cycle 1 Day 1 pre-dose and up to 24 hours post-dose
Population: This analysis was not performed due to lack of data.
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: AUC(Last): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration in Phase 1b for TAK-117
Time Frame: Cycle 1 Day 1 pre-dose and up to 24 hours post-dose
Population: This analysis was not performed due to lack of data.
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: CL/F: Oral Clearance for TAK-117
Time Frame: Cycle 1 Day 1 pre-dose and up to 24 hours post-dose
Population: This analysis was not performed due to lack of data.
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: T1/2: Terminal Phase Elimination Half-life (T1/2) for TAK-117
Time Frame: Cycle 1 Day 1 pre-dose and up to 24 hours post-dose
Population: This analysis was not performed due to lack of data.
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: TAK-117 Plasma Concentrations When Administered 1 Day After Docetaxel in Phase 2
Time Frame: 1 day post docetaxel dose
Population: Data was not analyzed as Phase 2 of study was cancelled.
Arm/Group | Phase 2 - TAK-117 + Docetaxel 36 mg/m^2 | Phase 2 - Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug through 30 days from the last dose (up to Day 223)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/6 | 3/8
Serious Adverse Events (participants affected / at risk) | 5/6 | 6/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 (N=6) | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2 (N=8)
Pneumonia (Infections and infestations) | 2 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Legionella infection (Infections and infestations) | 0 | 1 — One treatment-emergent death occurred during treatment with TAK-117 300 mg + Docetaxel and was not related.
Sepsis (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with TAK-117 300 mg + Docetaxel and was related.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with TAK-117 200 mg + Docetaxel and was not related.
Cardiogenic shock (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One treatment-emergent death occurred during treatment with TAK-117 300 mg + Docetaxel and was not related.
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - TAK-117 200 mg + Docetaxel 36 mg/m^2 (N=6) | Phase 1 - TAK-117 300 mg + Docetaxel 36 mg/m^2 (N=8)
Vision blurred (Eye disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fatigue (General disorders) | 3 | 4
Oedema peripheral (General disorders) | 2 | 2
Pyrexia (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT02393209/SAP_000.pdf
  • Study Protocol (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT02393209/Prot_001.pdf